CLINICAL TRIAL: NCT04417842
Title: CLOUD Study: Connect Lung Outcomes With Bronchodilator Use
Brief Title: Connect Lung Outcomes With Bronchodilator Use
Acronym: CLOUD
Status: Completed | Type: Observational
Sponsor: Pulmonary Critical Care Associates of Baltimore (Other)
Responsible Party: Principal Investigator, Alan Schwartz, Principal Investigator, Pulmonary Critical Care Associates of Baltimore
Other Study IDs: V1 21APR2020
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Respimetrix flow-volume monitoring device — The Respimetrix flow-volume monitoring device is being tested to validate its ability to measure Inspiratory Capacity

SUMMARY:
To determine the accuracy of the Respimetrix flow-volume monitoring device in measuring the patient's inspiratory capacity as compared to gold-standard measurements of inspiratory capacity on pulmonary function testing. Accuracy will be assessed before and after (A) pulmonary function testing and before and after (B) the administration of an inhaled bronchodilator medication.

DETAILED DESCRIPTION:
1. Specific Aim #1: Compare the performance of the flow-volume test device to standard pulmonary function measurements.

   The investigators hypothesize that measurements of inspiratory capacity with the Respimetrix test device will:

   A. Accurately measure the inspiratory capacity as assessed on standard pulmonary function tests, and will B. Correlate with other measures of pulmonary function including spirometry (vital capacity, forced expiratory volume in 1 second) and lung volumes (total lung capacity, functional residual capacity and residual volume).
2. Specific Aim #2: Examine the ability of the flow-volume test device to track changes in standard pulmonary function measurements after the administration of an inhaled bronchodilator.

The investigators hypothesize that the Respimetrix test device will:

A. Accurately measure changes in inspiratory capacity in response to a standard dose of a short acting inhaled beta-agonist (4 puffs albuterol), B. Correlate with immediate changes in pulmonary function parameters including spirometry (vital capacity, forced expiratory volume in 1 second) and lung volumes (total lung capacity, functional residual capacity and residual volume).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who are being seen in the pulmonary clinic including Asthma and Chronic Obstructive Pulmonary Disease (COPD) patients.
* Patients must be willing and able to provide informed consent to participate in the study.
* Patients must be able to use a metered dose inhaler.

Exclusion Criteria:

* Contraindication to inhaler use
* Tracheostomy
* Incapacitating disability that interferes with the use of the inhaler or execution of the protocol
* Unable to understand informed consent (e.g., non-English speakers)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Patients 18 years of age or older who are being seen in the pulmonary clinic including Asthma and COPD patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Validation | 1 year
  Validate the Respimetrix device as compared to pulmonary function test

SECONDARY OUTCOMES:
Validation | 1 year
  Validate Forced Vital Capacity, Forced expired volume in 1 sec, Total lung capacity and residual volume

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary and Critical Care Associates Of Baltimore, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Validating a device for Respimetrix, no immediate plan to share data.